CLINICAL TRIAL: NCT05972759
Title: Identifying the Neural Signature of Exercise to Advance Treatment of PD Cognitive Declines
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jay Alberts, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-568
Record Dates: First submitted 2023-07-11; First posted 2023-08-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; DBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Twenty-five participants with PD utilizing the Medtronic Percept PC DBS system will be enrolled for this project and completed a single bout of both FE and VE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Two modes of high intensity exercise.
  Interventions: Other: Forced and voluntary exercise

INTERVENTIONS:
Other: Forced and voluntary exercise — Twenty-five participants with PD utilizing the Medtronic Percept PC DBS system will be enrolled for this project and complete a single bout of both FE and VE. The 150-minute experimental session will be completed in the OFF antiparkinsonian and Off-DBS state.

SUMMARY:
Twenty-five participants with PD utilizing the Medtronic Percept PC DBS system will be enrolled for this project and complete a single bout of both FE and VE. The 150-minute experimental session will be completed in the OFF antiparkinsonian and Off-DBS state.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurological disease, most prevalent in older adults, estimated to affect over 12 million people world-wide by 2040. Traditionally considered a motor disorder, the impact of PD on cognitive performance is now widely accepted with 80% of PD patients developing executive function impairments. Typical PD related cognitive effects include impaired information processing, set-switching, working memory and dual-tasking. While antiparkinsonian medication and deep brain simulation (DBS) are effective in managing disease symptoms, disease modification has remained elusive. Exercise has been proposed as the Universal Prescription for PD capable of slowing disease progression; stationary cycling in particular has been suggested as an ideal exercise modality for people with PD (PwPD). The investigator's seminal tandem cycling study was the first to utilize forced exercise (FE) in human PD patients and demonstrated a 30% improvement in clinical ratings compared to voluntary exercise (VE). Briefly, FE is a mode of high intensity exercise originating in animal models of PD in which voluntary exercise rate is augmented, but not replaced. Thus, PwPD were assisted in pedaling at a higher rate (cadence) on the tandem cycle compared to those on a standard stationary cycle performing voluntary exercise (VE). This work resulted in a paradigm shift in terms of recommending high intensity exercise for PwPD. Despite the potential of exercise to alter disease progression, its mechanism of action and effects on basal ganglia function are not understood.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a diagnosis of PD by a movement disorders neurologist
* Previous placement, at least six months, of bilateral Medtronic Precept DBS as standard of care treatment for their PD.
* Stable and clinically optimized DBS parameters for three months prior to enrollment.
* Demonstrate the ability to safely mount and dismount a recumbent exercise cycle with an upright back.
* Willingness to withhold antiparkinsonian medication and DBS stimulation.
* Exercise clearance using the American College of Sports Medicine (ACSM) Pre-participation Health Screen: a. If the ACSM screen recommends medical clearance, the subject must obtain medical clearance by their health care provider prior to participation; b. Those who choose not to obtain physician clearance will not be eligible for participation.

Exclusion Criteria:

* Diagnosis of dementia or any neurocognitive impairment that compromises the ability to provide informed consent.
* A musculoskeletal issue that limits one's ability to cycle
* Neurological disease other than Parkinson's disease (i.e. multiple sclerosis, stroke) that impacts motor or cognitive function
* Uncontrolled cardiovascular risk factor such as a current cardiac arrhythmia, uncontrolled hypertension, untreated deep vein thrombosis, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Local Field Potentials during Cognitive Testing | an average of 3 total days
  Change in power in frequency bands of interest
Trail Making Test A & B | an average of 3 total days
  Change in neuropsychological tests designed to evaluate set-switching and attention
Information Processing | an average of 3 total days
  Change in mobile application of simple and choice reaction time
N-Back Test | an average of 3 total days
  Change in working memory test of word recall
Force-tracking with n-back | an average of 3 total days
  Change in upper extremity motor control assessment with cognitive component

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, Ph.D., Principal Investigator — Staff
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Koop MM, Rosenfeldt AB, Berki V, Bazyk A, Davidson S, Malan NS, Nagel S, Walter BL, Liao JY, Alberts JL. A novel methodological approach to understanding the cortical and subcortical effects of aerobic exercise in Parkinson's disease. Front Hum Neurosci. 2025 Oct 20;19:1657049. doi: 10.3389/fnhum.2025.1657049. eCollection 2025. PMID 41189627